CLINICAL TRIAL: NCT06422793
Title: The Impact of Nasogastric Tube Gastric Decompression on Postoperative Nausea and Vomiting in Orthognathic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Katherine Curry, Dr., Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1030776
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Nausea; Postoperative Vomiting
Keywords: nasogastric tube; orthognathic surgery; gastric decompression
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: This is a prospective study for patients undergoing orthognathic surgery at the Victoria General Hospital who meet study inclusion criteria. Participants are randomized into one of two study groups represented by no NG tube gastric decompression or NG tube gastric decompression intra-operatively and for one hour post-operatively. Participants are sequentially assigned to their study group using a randomized protocol list at the time of enrolment.
Who Masked: Participant
Masking Description: Participants will be blinded from their treatment group to minimize placebo effect, although they may later recall NG tube presence/removal if they belong in the NG group. Surgeons and anesthesiologists will not be blinded, as the nature of the study is not conducive to a double-blinded method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No NG Gastric Decompression (Experimental): No NG tube gastric decompression for orthognathic surgery. This group will not have a NG tube inserted. The remainder of their surgical care will be identical to the other group. PONV will be evaluated by nursing and surgical team at two time points in the 24 hour postoperative period (early [0-2 hours] and delayed [2-24 hours]).
  Interventions: Procedure: No NG tube gastric decompression
- NG Gastric Decompression (No Intervention): Participants will undergo NG tube gastric decompression according to our institution's typical gastric decompression regimen. Once patients are anesthetized and intubated, and a #14 French NG tube will be inserted in the naris opposite the nasotracheal tube and hooked up to low suction to confirm placement. If in the correct position, gastric contents will be seen in suction tubing. If no gastric contents are seen, the NG tube will be adjusted accordingly. The NG tube will be connected to suction until all stomach contents are effectively removed, as demonstrated by no new secretions in the suction tubing. It will then be disconnected from suction, secured with tape throughout surgery and temporarily hooked back up to suction at the end of surgery to reconfirm position and suction stomach contents present. The NG tube will then be secured and left in place for one hour on intermittent suction following arrival to the recovery unit. After one hour, the NG tube will be removed.

INTERVENTIONS:
Procedure: No NG tube gastric decompression — Participants in this group will not undergo gastric decompression following orthognathic surgery at our institution.
  Arms: No NG Gastric Decompression

SUMMARY:
This study will compare the incidence of postoperative nausea and vomiting during the first 24 hours following corrective jaw surgery (orthognathic surgery) in patients with and without nasogastric tube gastric decompression.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) affects up to 60% of patients after orthognathic surgery. Multiple complex mechanisms contribute to the development of PONV, but gastric pooling of blood is speculated to be the primary stimulus in this type of surgery. Nasogastric (NG) tubes can be used for gastric decompression in the peri-operative period to evacuate gastric contents/blood, with an intent to minimize PONV. This study will directly compare the incidence of PONV in participants undergoing NG tube gastric decompression and those without NG tube gastric decompression in the first 24 hours after orthognathic surgery. Participants will be randomized into two groups including no NG tube gastric decompression or NG tube gastric decompression throughout the surgery with removal one one hour postoperatively. The presence of early and/or delayed PONV will be monitored to determine the impact of NG tube gastric decompression. This study will also evaluate the impact of other variables including type of anesthesia, length of surgery, type of surgery and patient factors on the incidence of PONV in this study population.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 16 at the time of consent undergoing orthognathic surgery for the correction of dentofacial deformities at the Victoria General Hospital during the study period.

Orthognathic surgery to include:

1. Patients who receive single-jaw surgery (i.e. BSSO [Bilateral Sagittal Split Osteotomy] only, or LeFort only).
2. Patients receiving double-jaw surgery (i.e. BSSO and LeFort).
3. Patients undergoing a functional genioplasty in addition to another osteotomy (i.e. BSSO and/or LeFort).

Exclusion Criteria:

* Patients will be excluded if they do not meet inclusion criteria or if they have risk factors known to directly impact PONV and/or cause delayed gastric emptying:

  1. Patients under the age of 16 at the time of consent.
  2. Patients contraindicated to undergo elective surgery, including pregnant patients.
  3. Patients undergoing a functional genioplasty procedure only.
  4. Patients taking GLP-1 receptor agonists).
  5. Patients with known gastroparesis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting | Participants will be assessed for early PONV (0-2 hours postoperatively) and delayed PONV (2-24 hours postoperatively).
  The primary outcome for this study is PONV characterized by nausea and/or emesis in participants subject to one of two NG tube gastric decompression protocols during the 24-hour postoperative period. This will be characterized by indicating presence of nausea or vomiting with "yes" or "no" at two different time points (early vs delayed PONV).

SECONDARY OUTCOMES:
NG Tube Related Complications/Factors | Intraoperative documentation during NG tube insertion.
  Evaluating factors related to NG tubes including the incidence of NG tube-related complications and the length of time taken to successfully insert a NG tube. Any complications will be documented. Length of time taken to insert the tube will be recorded in seconds. This data will be described using percent for incidence and descriptive statistics.
Incidence of Early vs Delayed PONV in our Study Population | Participants will be assessed for early PONV (0-2 hours postoperatively) and delayed PONV (2-24 hours postoperatively).
  Evaluate whether participants tend to experience more early (0-2h) or delayed (2-24h) PONV, increasing our understanding of possible precipitants. This will be characterized by indicating presence of nausea or vomiting with "yes" or "no" at two different time points (early [0-2 hours postoperatively] vs delayed [2-24 hours postoperatively]).
Other Factors Impacting PONV | Participants will be assessed for early PONV (0-2 hours postoperatively) and delayed PONV (2-24 hours postoperatively).
  Gain better understanding how patient demographics, length of surgery, type of surgery, and type of general anesthesia impact PONV in our study population. Participant's age (years), sex (male or female), smoking status (smoker or non-smoker), history of PONV or motion sickness (positive or negative), length of surgery (from first incision to closure), type of orthognathic surgery (LeFort, BSSO, or both), type of general anesthesia (total intravenous anesthetic vs combined volatile/ intravenous anesthetic) will be evaluated for correlation to PONV in the 24 hour postoperative period.
Apfel Score as a Predictor of PONV in our Study Population | Apfel score will be determined preoperatively. Participants will be assessed for early PONV (0-2 hours postoperatively) and delayed PONV (2-24 hours postoperatively).
  Evaluating whether Apfel scores correlate to PONV and can function as an accurate predictor of PONV in our study population.The Apfel score (0-4) will be documented for each patient. Apfel score means for groups experiencing nausea and/or vomiting will be compared to Apfel score means for participants who do not experience nausea and/or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: James Brady, DDS/MD, Principal Investigator — NSHA
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
This data will be anonymous. Participants will only be consenting to participate in this study. There is no future studies planned using this study data.

REFERENCES:
- [Background] Koivuranta M, Laara E, Snare L, Alahuhta S. A survey of postoperative nausea and vomiting. Anaesthesia. 1997 May;52(5):443-9. doi: 10.1111/j.1365-2044.1997.117-az0113.x. PMID 9165963
- [Background] Becker DE. Nausea, vomiting, and hiccups: a review of mechanisms and treatment. Anesth Prog. 2010 Winter;57(4):150-6; quiz 157. doi: 10.2344/0003-3006-57.4.150. PMID 21174569
- [Background] Ghosh S, Rai KK, Shivakumar HR, Upasi AP, Naik VG, Bharat A. Incidence and risk factors for postoperative nausea and vomiting in orthognathic surgery: a 10-year retrospective study. J Korean Assoc Oral Maxillofac Surg. 2020 Apr 30;46(2):116-124. doi: 10.5125/jkaoms.2020.46.2.116. PMID 32364351
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Kovac AL. Prevention and treatment of postoperative nausea and vomiting. Drugs. 2000 Feb;59(2):213-43. doi: 10.2165/00003495-200059020-00005. PMID 10730546
- [Background] Apipan B, Rummasak D, Wongsirichat N. Postoperative nausea and vomiting after general anesthesia for oral and maxillofacial surgery. J Dent Anesth Pain Med. 2016 Dec;16(4):273-281. doi: 10.17245/jdapm.2016.16.4.273. Epub 2016 Dec 31. PMID 28879315
- [Background] Zhong W, Shahbaz O, Teskey G, Beever A, Kachour N, Venketaraman V, Darmani NA. Mechanisms of Nausea and Vomiting: Current Knowledge and Recent Advances in Intracellular Emetic Signaling Systems. Int J Mol Sci. 2021 May 28;22(11):5797. doi: 10.3390/ijms22115797. PMID 34071460
- [Background] Dobbeleir M, De Coster J, Coucke W, Politis C. Postoperative nausea and vomiting after oral and maxillofacial surgery: a prospective study. Int J Oral Maxillofac Surg. 2018 Jun;47(6):721-725. doi: 10.1016/j.ijom.2017.11.018. Epub 2018 Jan 1. PMID 29301675
- [Background] Silva AC, O'Ryan F, Poor DB. Postoperative nausea and vomiting (PONV) after orthognathic surgery: a retrospective study and literature review. J Oral Maxillofac Surg. 2006 Sep;64(9):1385-97. doi: 10.1016/j.joms.2006.05.024. PMID 16916674
- [Background] Apfel CC, Roewer N. Risk assessment of postoperative nausea and vomiting. Int Anesthesiol Clin. 2003 Fall;41(4):13-32. doi: 10.1097/00004311-200341040-00004. No abstract available. PMID 14574212
- [Background] Laskin DM, Carrico CK, Wood J. Predicting postoperative nausea and vomiting in patients undergoing oral and maxillofacial surgery. Int J Oral Maxillofac Surg. 2020 Jan;49(1):22-27. doi: 10.1016/j.ijom.2019.06.016. Epub 2019 Jun 21. PMID 31230771
- [Background] Pourtaheri N, Peck CJ, Maniskas S, Park KE, Allam O, Chandler L, Smetona J, Yang J, Wilson A, Dinis J, Lopez J, Steinbacher DM. A Comprehensive Single-Center Analysis of Postoperative Nausea and Vomiting Following Orthognathic Surgery. J Craniofac Surg. 2022 Mar-Apr 01;33(2):584-587. doi: 10.1097/SCS.0000000000008052. PMID 34510064
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Sanaie S, Mahmoodpoor A, Najafi M. Nasogastric tube insertion in anaesthetized patients: a comprehensive review. Anaesthesiol Intensive Ther. 2017;49(1):57-65. doi: 10.5603/AIT.a2017.0001. Epub 2017 Jan 13. PMID 28084614
- [Background] Kerger KH, Mascha E, Steinbrecher B, Frietsch T, Radke OC, Stoecklein K, Frenkel C, Fritz G, Danner K, Turan A, Apfel CC; IMPACT Investigators. Routine use of nasogastric tubes does not reduce postoperative nausea and vomiting. Anesth Analg. 2009 Sep;109(3):768-73. doi: 10.1213/ane.0b013e3181aed43b. PMID 19690245
- [Background] Wang J, Zhang Z. Gastric Negative Pressure Suction Method Reduces the Incidence of PONV after Orthognathic Surgery. Front Surg. 2022 May 20;9:882726. doi: 10.3389/fsurg.2022.882726. eCollection 2022. PMID 35669253
- [Background] Schmitt ARM, Ritto FG, de Azevedo JGRL, Medeiros PJD, de Mesquita MCM. Efficacy of Gastric Aspiration in Reducing Postoperative Nausea and Vomiting After Orthognathic Surgery: A Double-Blind Prospective Study. J Oral Maxillofac Surg. 2017 Apr;75(4):701-708. doi: 10.1016/j.joms.2016.10.002. Epub 2016 Oct 12. PMID 27816732
- [Background] Maza, C., López, A. M., Kulyapina, A., Leno, B., Tousidonis, M., Garcia, A. & Salmerón, J. I. (2013). Orthognathic surgery: nasogastric tube responsible of the nausea and vomiting?. International Journal of Oral and Maxillofacial Surgery, 42(10), 1333.